CLINICAL TRIAL: NCT03259438
Title: Testing the Effects of Movement Based Interventions on Brain-Body Mechanisms in Fatigued Cancer Survivors
Brief Title: The Vitality Project for Fatigued Female Cancer Survivors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Miriam Hospital (Other)
Collaborators: Brown University (Other)
Responsible Party: Principal Investigator, Ellen Flynn, MD, Psychiatry, The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MiriamH 1040485
Record Dates: First submitted 2017-07-19; First posted 2017-08-23 (Actual); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Fatigue; Cancer Survivorship
Keywords: Qigong; Comprehensive Health Improvement Program (CHIP); Pre-Train Injury Prevention Program; Cancer Related Fatigue; Cancer Survivorship; Inflammation; Flowmetry; Corticomuscular coherence; Heart Rate Variability; Neuroimmune Interactions; Complex Systems Analysis; Female
MeSH Terms: conditions — Fatigue; Inflammation | interventions — Qigong; Chromatin Immunoprecipitation Sequencing

STUDY DESIGN:
Intervention Model Description: This parallel, randomized non-inferiority trial will test whether qigong is not inferior to an exercise/nutrition active comparator group in terms of reducing fatigue in female cancer survivors. If non-inferiority is demonstrated during analysis, a secondary analysis will test whether qigong can be considered superior to the exercise-nutrition comparator
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants will not find out what interventional group they are placed in (qigong vs. healthy living) until after they have completed their first testing session.
  Pre intervention data collection and post intervention data analysis will be completely masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Qigong (Experimental): This course will meet twice weekly for 2 hours and 15 minutes per class for ten weeks. Topics will include guided instruction in the theory and background of qigong and healing. Practice will include gentle stretching and guided qigong movement as well as seated and lying down meditations. Participants will be asked to complete about 30 minutes a day of home assignments.
  Interventions: Behavioral: Qigong
- Healthy Living (CHIP + Pre-Train) (Active Comparator): This course will meet twice weekly for 2 hours and 15 minutes per class for ten weeks. Topics will include plant based nutrition counseling via the Comprehensive Health Improvement Program (CHIP) as well as core-stretching, strengthening, and light aerobic movements through a Pre-Train exercise program. Participants will be asked to complete about 30 minutes a day of home assignments.
  Interventions: Behavioral: Healthy Living (CHIP + Pre-Train)

INTERVENTIONS:
Behavioral: Qigong — Qigong is a form of gentle mind-body movement that originates in China and has traditionally been used for healing purposes. It has been reported to improve energy levels, as well as strength and endurance and mental clarity and equanimity. This study will assess how a 10-week qigong intervention compares to an exercise-nutrition intervention in improving fatigue and vitality in female cancer survivors. On a secondary level, we will asses changes in underlying brain, heart, and peripheral dynamics that occur as a result of the qigong practice to develop a mechanistic understanding of qigong's efficacy.
  Arms: Qigong
Behavioral: Healthy Living (CHIP + Pre-Train) — The Healthy Living active comparator intervention includes two components: plant based nutrition counseling via the Comprehensive Health Improvement Program (CHIP) and core strengthening exercises and light aerobic activity via the Pre-Train exercise program.
  Arms: Healthy Living (CHIP + Pre-Train)

SUMMARY:
This parallel, randomized, non-inferiority trial will examine whether a ten week qigong intervention is not inferior to a ten week exercise-nutrition comparison group in reducing fatigue in cancer survivors. To build a more mechanistic understanding of physiological changes associated with fatigue reduction, it will secondly collect several different types of data to build an integrative brain-body model of vigor in cancer survivorship including:

1. data related to neural correlates of body awareness: cortical EEG data measuring each subject's ability to use attention to control neurons in primary somatosensory cortex (replication of Kerr et al 2011 study in mindfulness), and resting state fMRI measures of insular connectivity with nodes of the default mode network and salience network
2. data related to inflammation measured via inflammatory cytokines (e.g., interleukin-6 and tnf-alpha)
3. data related to cardiorespiratory functioning including cardiac impedance (ICG) and mechanical lung function
4. data related to parasympathetic and sympathetic signaling between the nervous system and the rest of the periphery.

DETAILED DESCRIPTION:
The purpose of this study is to examine the therapeutic effects of movement and body awareness on recovery from cancer-related fatigue. In the current study, 60-80 female cancer survivors with cancer-related fatigue will be recruited who have been out of treatment for at least eight weeks. They will be randomized to either a 10-week qigong contemplative movement course or a 10 -week exercise-nutrition course. This study is designed as a non-inferiority trial to test the primary hypothesis that a ten week qigong intervention is not inferior to a ten week exercise-nutrition active comparator group in reducing fatigue in female cancer survivors (assessed via the FACIT-Fatigue scale). If non-inferiority is demonstrated during analysis, the data will be further analyzed to examine whether the qigong group significantly decreases fatigue more than the healthy living comparison group. The FACIT-Fatigue scale will be delivered at three time points: before the intervention starts (T1), after it ends (T2), and three months after the intervention has ended (T3). Further, this study will directly examine the underlying physiological mechanisms by which each intervention exerts its effects. Participants will be tested pre (T1) and post (T2) intervention on a variety of measures across multiple bodily and brain systems (eg EEG, fMRI, EMG, ECG, ICG, mechanical lung function, Doppler flowmetry, serum cytokines, muscle strength, 6 min walk test) to assess changes in these systems that are associated with reduction of fatigue and improvement of the subjective sense of vitality and energy. The data will be used to test whether conscious attention to bodily sensations cultivated in contemplative movement practices (i.e. Qigong) can actually impact levels of inflammation in the periphery as well as cortical measures of interoceptive awareness (ie resting state insula connectivity), and whether these changes will be associated with fatigue reduction. The secondary hypothesis is that decreased inflammation levels in the blood will be correlated with reduction in fatigue at post intervention as well as changes in neural markers of interoceptive and bodily awareness, and that this effect will be stronger in the qigong group.

ELIGIBILITY:
Inclusion Criteria:

* Female patients
* Aged 18-70 years
* Have completed a course of chemotherapy cancer treatment (except for ongoing treatment with Herceptin [trastuzumab] or other adjuvant therapies), AND/OR radiation treatment, AND/OR surgery, with no surgery, radiation or chemotherapy received in the past 8 weeks.
* Endorse a 3/10 or above for the question "On a scale of one to ten, in the last week, how much has your fatigue interfered with your daily life, with 1 being not at all, and 10 being all the time" AND/OR "On a scale of one to ten, in the last week, how much have you felt your sleep has been disturbed or of a quality that you have not felt rested when you wake up, with 1 being not at all, and 10 being all the time"
* Have a primary care or other physician
* Ability to understand English
* Willingness to have blood drawn
* Willingness to have an EEG, EKG, and EMG taken
* Willingness to complete questionnaires
* Willingness and ability to undergo an fMRI scan (screening parameters for this are included below) [optional: participant doesn't have to do this if it will represent too much burden to the participant, or if they have other contraindications to fMRI such as metal in the body, etc.]
* Ability to pass basic validated physical movement tests (e.g.: standing with feet touching for 30 seconds, twist right to left and back, hold arms out to side in air for 15 seconds, lift arms over head, moving from standing position to seated position on the floor) to verify safety for qigong and exercise practices

Exclusion Criteria:

* History or current diagnosis of coronary artery or coronary heart disease
* History or current diagnosis of heart attack, or heart murmur
* Electrical Pacemaker Implant in heart
* Peripheral neuropathy in hands
* History or current diagnosis of any other MAJOR psychiatric disorder (including psychosis, or mania, or suicidal or homicidal ideation) besides depression or anxiety
* Active alcohol or drug abuse
* Tobacco use
* Pregnancy
* Ingestion of caffeine or cocoa products less than two hours from data collection
* Inability to participate in gentle exercises (like pilates)

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Must be female
Enrollment: 75 (Estimated)
Dates: Start 2017-07-24 (Actual); Primary Completion 2017-12-20 (Estimated); Study Completion 2018-01-30 (Estimated)

PRIMARY OUTCOMES:
Reduction in Fatigue (via FACIT-Fatigue scale) | Measured at baseline (time 1) and after 10-week intervention (time 2) and 3 months after end of intervention (time 3)
  Fatigue assessed via the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) questionnaire

SECONDARY OUTCOMES:
Electrocardiogram (ECG) | Measured at baseline (time 1) and after 10-week intervention (time 2)
  Will be measured to calculate heart rate variability (HRV)
Impedance Cardiography | Measured at baseline (time 1) and after 10-week intervention (time 2)
  Will be used to assess exercise related improvements in cardiovascular tone.
Electroencephalography (EEG) | Measured at baseline (time 1) and after 10-week intervention (time 2)
  Will be used to assess changes in cortical brain waves (particularly alpha and beta rhythms)
Tactile Acuity | Measured at baseline (time 1) and after 10-week intervention (time 2)
  A task that involves subtle taps to the finger tips, EEG is simultaneously recorded to examine modulation in brain rhythms across somatosensory cortex related to cued attention to the tap
Electromyography (EMG) | Measured at baseline (time 1) and after 10-week intervention (time 2)
  A measure of muscle rhythms
Precision Grip | Measured at baseline (time 1) and after 10-week intervention (time 2)
  A measure of one's ability to hold a lever at a steady force, EEG and EMG simultaneously record corticomuscular coherence that may facilitate steady grip
Electrodermal Activity (skin conductance) | Measured at baseline (time 1) and after 10-week intervention (time 2)
  to assess sympathetic tone
Working memory capacity (WMC) | Measured at baseline (time 1) and after 10-week intervention (time 2)
  Assessed via the short-form O-SPAN computer-based task to assess overall memory impairments
Mechanical lung function | Measured at baseline (time 1) and after 10-week intervention (time 2)
  to determine the impact of exercise and movement on overall lung function
Inflammatory cytokines (eg Il-1, Il-6) collected via a blood draw | Measured at baseline (time 1) and after 10-week intervention (time 2)
  To measure the interaction between the brain measures of bodily awareness and the immune system
Resting State Functional Magnetic Resonance Imaging (rs-fMRI) | Measured at baseline (time 1) and after 10-week intervention (time 2)
  Optional measure: To assess changes in functional connectivity associated with participation in the intervention
Muscle Strength | Measured at baseline (time 1) and after 10-week intervention (time 2)
  Assessed via jamar hand dynamometers and back, leg, and arm dynamometers to assess changes in muscle tone associated with the classes
6 Minute Walk Test | Measured at baseline (time 1) and after 10-week intervention (time 2)
  Test of how far a participant can walk in six minutes to assess overall endurance
Patient Health Questionnaire | Measured at baseline (time 1) and after 10-week intervention (time 2) and 3 months after end of intervention (time 3)
  Measure of anxiety and depression
Functional Assessment of cancer therapy-General (FACT-G) Questionnaire | Measured at baseline (time 1) and after 10-week intervention (time 2) and 3 months after end of intervention (time 3)
  Measure of physical, social, emotional, and functional well-being
Multidimensional Assessment of Interoceptive Awareness (MAIA) Questionnaire | Measured at baseline (time 1) and after 10-week intervention (time 2) and 3 months after end of intervention (time 3)
  Questionnaire to measure subjectively reported interoceptive and bodily awareness (including body-specific sensations, emotions, and cognitions)
Profile of Mood States (POMS) Questionnaire | Measured at baseline (time 1) and after 10-week intervention (time 2) and 3 months after end of intervention (time 3)
  To assess fatigue, vigor, and overall mood
Pittsburgh Sleep Quality Index (PSQI) | Measured at baseline (time 1) and after 10-week intervention (time 2) and 3 months after end of intervention (time 3)
  Measurement of sleep quality, habits, and patterns
Rand 36-Item Short Form Health Survey (SF-36) | Measured at baseline (time 1) and after 10-week intervention (time 2) and 3 months after end of intervention (time 3)
  Measurement of overall quality of life
Difficulties in Emotion Regulation Scale (DERS) | Measured at baseline (time 1) and after 10-week intervention (time 2) and 3 months after end of intervention (time 3)
  Measures multiple factors of emotional dysregulation
Fatigue Symptom Inventory (FSI) | Measured at baseline (time 1) and after 10-week intervention (time 2) and 3 months after end of intervention (time 3)
  Measures overall fatigue interfrerence

OTHER OUTCOMES:
Apple watches Heart Rate and Physical Steps Tracking | Optional Measure: For those involved, tracked daily for five days before the intervention starts, for the 70 days during the 10-week intervention, and for five days after the intervention ends.
  Apple watches will be supplied to interested participants to monitor their heart rate and physical steps taken throughout the day to assess changes in movement patterns while participating in the classes
Perceived Stress Scale (PSS) Questionnaire | Measured at baseline (time 1) and after 10-week intervention (time 2) and 3 months after end of intervention (time 3)
  To assess changes in self-reported stress
Multidimensional Scale of Perceived Social Support (MSPSS) | Measured at baseline (time 1) and after 10-week intervention (time 2) and 3 months after end of intervention (time 3)
  Measure of self-reported social support
Unmitigated Communion Scale | Measured at baseline (time 1) and after 10-week intervention (time 2) and 3 months after end of intervention (time 3)
  A measure of a person's tendency to care for other's before themselves
Godin Leisure time Questionnaire | Measured at baseline (time 1) and after 10-week intervention (time 2) and 3 months after end of intervention (time 3)
  Measure of how much a person has been excising or relaxing

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Flynn, MD, Principal Investigator — The Miriam Hospital
Locations (1):
- Miriam Hospital Outpatient 146 West River Street, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No
No sharing plan anticipated.

REFERENCES:
- [Background] Farb N, Daubenmier J, Price CJ, Gard T, Kerr C, Dunn BD, Klein AC, Paulus MP, Mehling WE. Interoception, contemplative practice, and health. Front Psychol. 2015 Jun 9;6:763. doi: 10.3389/fpsyg.2015.00763. eCollection 2015. PMID 26106345
- [Background] Desbordes G, Gard T, Hoge EA, Holzel BK, Kerr C, Lazar SW, Olendzki A, Vago DR. Moving beyond Mindfulness: Defining Equanimity as an Outcome Measure in Meditation and Contemplative Research. Mindfulness (N Y). 2014 Jan 21;2014(January):356-72. doi: 10.1007/s12671-013-0269-8. PMID 25750687
- [Background] Wells RE, Yeh GY, Kerr CE, Wolkin J, Davis RB, Tan Y, Spaeth R, Wall RB, Walsh J, Kaptchuk TJ, Press D, Phillips RS, Kong J. Meditation's impact on default mode network and hippocampus in mild cognitive impairment: a pilot study. Neurosci Lett. 2013 Nov 27;556:15-9. doi: 10.1016/j.neulet.2013.10.001. Epub 2013 Oct 10. PMID 24120430
- [Background] Daubenmier J, Sze J, Kerr CE, Kemeny ME, Mehling W. Follow your breath: respiratory interoceptive accuracy in experienced meditators. Psychophysiology. 2013 Aug;50(8):777-89. doi: 10.1111/psyp.12057. Epub 2013 May 22. PMID 23692525
- [Background] Kerr CE, Sacchet MD, Lazar SW, Moore CI, Jones SR. Mindfulness starts with the body: somatosensory attention and top-down modulation of cortical alpha rhythms in mindfulness meditation. Front Hum Neurosci. 2013 Feb 13;7:12. doi: 10.3389/fnhum.2013.00012. eCollection 2013. PMID 23408771
- [Background] Kerr CE, Jones SR, Wan Q, Pritchett DL, Wasserman RH, Wexler A, Villanueva JJ, Shaw JR, Lazar SW, Kaptchuk TJ, Littenberg R, Hamalainen MS, Moore CI. Effects of mindfulness meditation training on anticipatory alpha modulation in primary somatosensory cortex. Brain Res Bull. 2011 May 30;85(3-4):96-103. doi: 10.1016/j.brainresbull.2011.03.026. Epub 2011 Apr 8. PMID 21501665
- [Background] Mehling WE, Wrubel J, Daubenmier JJ, Price CJ, Kerr CE, Silow T, Gopisetty V, Stewart AL. Body Awareness: a phenomenological inquiry into the common ground of mind-body therapies. Philos Ethics Humanit Med. 2011 Apr 7;6:6. doi: 10.1186/1747-5341-6-6. PMID 21473781
- [Background] Kerr CE, Shaw JR, Wasserman RH, Chen VW, Kanojia A, Bayer T, Kelley JM. Tactile acuity in experienced Tai Chi practitioners: evidence for use dependent plasticity as an effect of sensory-attentional training. Exp Brain Res. 2008 Jun;188(2):317-22. doi: 10.1007/s00221-008-1409-6. Epub 2008 May 30. PMID 18512052
- [Background] Lazar SW, Kerr CE, Wasserman RH, Gray JR, Greve DN, Treadway MT, McGarvey M, Quinn BT, Dusek JA, Benson H, Rauch SL, Moore CI, Fischl B. Meditation experience is associated with increased cortical thickness. Neuroreport. 2005 Nov 28;16(17):1893-7. doi: 10.1097/01.wnr.0000186598.66243.19. PMID 16272874
- [Derived] Zimmerman CS, Temereanca S, Daniels D, Penner C, Cannonier T, Jones SR, Kerr C. A Randomized Controlled Pilot Trial Comparing Effects of Qigong and Exercise/Nutrition Training on Fatigue and Other Outcomes in Female Cancer Survivors. Integr Cancer Ther. 2023 Jan-Dec;22:15347354231162584. doi: 10.1177/15347354231162584. PMID 37204076